CLINICAL TRIAL: NCT02912338
Title: The Effectiveness of Lifestyle Intervention on Body Composition, Physical Performances and Quality of Life Among Elderly People in Long-term Care Facilities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Taiwan University of Science and Technology (Other)
Responsible Party: Principal Investigator, Chiu Shu-Ching, Senior Lecturer, PhD candidate, Central Taiwan University of Science and Technology
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CTU104-PC-014
Record Dates: First submitted 2016-09-09; First posted 2016-09-23 (Estimated); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: Sarcopenia; Obesity
Keywords: Sarcopenic obesity; Body composition; Physical function; quality of life; long term care
MeSH Terms: conditions — Sarcopenia; Obesity | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Resistant Training Group (Experimental): sandbag 2-5lb, grip ball, twice/week, Duration:12 weeks
  Interventions: Behavioral: Resistant Training
- Control Group (Active Comparator): not change lifestyle
  Interventions: Other: Control Group

INTERVENTIONS:
Behavioral: Resistant Training
  Arms: Resistant Training Group
Other: Control Group
  Arms: Control Group

SUMMARY:
Purpose: To understand the change in body composition, physical functions and quality of life of elderly residents with sarcopenic obesity in LTC facilities after the implementation of exercise intervention.

ELIGIBILITY:
Inclusion Criteria:

1. aged and elderly over 60 years old and no exercise restrictions.
2. conscious clear, able to communicate with to the traditional Chinese language or Taiwanese.
3. in the past three months living in long-term care institutions.
4. in the last month the subject biased static life
5. in a stable condition with enough energy: to maintain the support of at least one hour sitting in a wheelchair or bed edge.

Exclusion Criteria:

1. In the past three months have unstable weight (> ± 4 kg).
2. severe disease states, such as severe heart and lung liver and kidney disease, a serious cancer, severe malnutrition (Mini Nutritional Assessment Scale 0-7 points).
3. limb unable to anti-gravity completely
4. severe dementia (Clinical Dementia Rating (CDR) Scale Clinical Dementia Rating, CDR 3-5 points).

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2015-09; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Body Composition | Change gram, kg and percentage from baseline to follow up (12 weeks later)
  measuring machine: Bioelectrical impedance analysis (BIA) estimates body composition of fat and lean tissue.
body weight | Change kg from baseline to follow up (12 weeks later)
  Weighing scales in kilograms
BMI | Change from baseline to follow up (12 weeks later)
  kg/m2
hand grip | Change from baseline to follow up (12 weeks later)
  Jamar Handgrip Dynamometer
hand pinch | Change kg from baseline to follow up (12 weeks later)
  Lafayette Hydraulic Pinch Gauge 5030P1
Activities of daily living | Change score from baseline to follow up (12 weeks later)
  Functional Independence Measure (FIM) included 18 items, covering 6 situations in the burden of personal care, specifically self-care, mobility, transfers, sphincter management, communication, and social cognition. A high score indicates better function.
Quality of Life | Change score from baseline to follow up (12 weeks later)
  Short Form 8 health survey (SF8)included the items focusing on physical and mental health; EuroQol-5D (EQ-5D) includes the EQ-visual analogue scale (VAS) and the EQ-5D descriptive system. EQ-VAS documents the participant's self-reported health on a VAS of 100-0. The EQ-5D-3L descriptive system consists of five dimensions, namely mobility, self-care, usual activities, pain/discomfort and anxiety/depression, all with three function levels (no problem = 1; some problems = 2; severe problems = 3)

REFERENCES:
- [Derived] Chang SF, Chiu SC. Effect of resistance training on quality of life in older people with sarcopenic obesity living in long-term care institutions: A quasi-experimental study. J Clin Nurs. 2020 Jul;29(13-14):2544-2556. doi: 10.1111/jocn.15277. Epub 2020 Apr 24. PMID 32279360
- [Derived] Chiu SC, Yang RS, Yang RJ, Chang SF. Effects of resistance training on body composition and functional capacity among sarcopenic obese residents in long-term care facilities: a preliminary study. BMC Geriatr. 2018 Jan 22;18(1):21. doi: 10.1186/s12877-018-0714-6. PMID 29357826